CLINICAL TRIAL: NCT03291405
Title: Correlation Between Body Mass Index and Gonadotrophin Secretions in Pcos Patients and Their Effect on Ivf Outcome (Randamized Control Trial)
Brief Title: Correlation Between Body Mass Index and Gonadotrophin Secretions in Pcos Patients and Their Effect on Ivf Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mahmoud sobhy, Correlation Between Body Mass Index and Gonadotrophin Secretions in Pcos Patients and Their Effect on Ivf Outcome, Ain Shams University
Other Study IDs: mahmoud
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Correlation Between Body Mass Index and Gonadotrophin Secretions in Pcos Patients and Their Effect on Ivf Outcome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Body Mass Index less than 30
- Body Mass Index more than 30

SUMMARY:
It is Correlation Between Body Mass Index and Gonadotrophin Secretions in Pcos Patients and Their Effect on Ivf Outcome

ELIGIBILITY:
Inclusion Criteria:

* cases of PCO

Exclusion Criteria:

* amenorrhea
* womenwho had previous IVF

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: total of 142 women will be involved
Sampling Method: Probability Sample
Enrollment: 142 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-02 (Estimated)

PRIMARY OUTCOMES:
Gonadotrophin Secretions in both groups | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt